CLINICAL TRIAL: NCT04162964
Title: Effectiveness of a Virtual Chair Yoga Intervention for Reducing Stress in Older Adults With Dementia and Caregivers
Brief Title: Chair Yoga for Stress in Dementia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: Lady Davis Institute (Other)
Responsible Party: Principal Investigator, Soham Rej MD, MSc, Principal Investigator, Lady Davis Institute
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GeriPARTy
Record Dates: First submitted 2019-10-29; First posted 2019-11-14 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2020-09

CONDITIONS: Dementia; Stress
Keywords: Dementia; Stress; Caregiving; Mind-body therapy; Anxiety; Depression
MeSH Terms: conditions — Dementia; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chair Yoga Treatment (Experimental)
  Interventions: Behavioral: Virtual Chair Yoga
- Waitlist Control Group (Placebo Comparator)
  Interventions: Behavioral: Virtual Chair Yoga

INTERVENTIONS:
Behavioral: Virtual Chair Yoga — 8-week virtual chair yoga program for one hour per week. Chair yoga is an effective way to offer modified yoga postures and relaxation techniques to individuals with limited mobility and/or advanced age for whom mat-based classes may not be accessible. The weekly yoga classes will be lead on the software Zoom by a certified instructor in English and French.

SUMMARY:
Over 700,000 Canadians are affected by dementia costing the health care system approximately $10 billion/year. Due to COVID-19, the government has urged individuals over the age of 70 to stay home, putting this population at risk of social isolation. Older adults with mild cognitive impairments (MCIs), dementia, and their caregivers are at an even higher risk of becoming stressed, anxious, and agitated while in lockdown. Unsurprisingly, caregiver burden is extremely common, and often precedes institutionalization of the patient, as the demands of the illness begin to exceed that which the caregiver can sustainably provide. Since social distancing measures have shut down activities and support groups for these individuals, there is an urgent need for scalable, cost-effective, non-pharmacological interventions that can be delivered remotely to improve stress and loneliness. Yoga may be a viable therapeutic modality to address the psychological challenges associated with dementia in patients and caregivers, as it has been shown to decrease stress and improve anxiety and depressive symptoms in various populations. For this reason, we are conducting a randomized controlled trial (RCT) to assess the efficacy of an 8-week virtual chair yoga program to improve stress, psychological symptoms, and caregiver burden. This virtual chair yoga study will engage both older adults with dementia/MCI and caregivers (n=40-60 participants) during COVID-19, which is consistent with the need for decreasing costs and increasing accessibility of novel health interventions during and beyond the pandemic. We will evaluate the effect of this program on stress, loneliness, and mental health related outcomes such as fear of COVID-19, depression, anxiety, and caregiver burden compared to a waitlist control group. We will also be conducting a qualitative component in the form of semi-structured interviews. All quantitative outcomes will be assessed before the program starts and post-intervention and qualitative outcomes will be assessed post-intervention. Participants will be randomly assigned to the treatment group (virtual chair yoga 1 hour per week on Zoom) or the waitlist control group. The investigators hypothesize that after the 8-week yoga program, older adults and caregivers will report lower stress, loneliness, depression, anxiety, fear of COVID-19, and caregiver burden. Results will be available late-2021.

ELIGIBILITY:
Inclusion Criteria for Older Adults:

* Mild cognitive impairment or mild to moderate dementia (MoCA-BLIND score between 8-18 OR a diagnosis from his/her clinician of mild cognitive impairment) or mild to moderate dementia
* Sufficient hearing to follow verbal instructions
* Access to Zoom software and internet connection
* Ability to sit for 60 minutes without discomfort
* At least 60 years old

Exclusion Criteria for Older Adults:

* Severe dementia (MoCA-BLIND score < 8)
* Acute psychotic symptoms
* Acute suicidal ideation or intent
* Resides outside of Quebec

Inclusion Criteria for Caregivers:

* Providing care for someone with cognitive impairments (mild cognitive impairment or mild, moderate, or severe dementia)
* Sufficient hearing to follow verbal instructions
* Access to Zoom software and internet connection
* Ability to sit for 60 minutes without discomfort
* At least 18 years old

Exclusion Criteria for Caregivers:

* Dementia (MoCA-BLIND score < 18)
* Acute psychotic symptoms
* Acute suicidal ideation or intent
* Resides outside of Quebec

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2021-03-13 (Actual); Study Completion 2021-03-13 (Actual)

PRIMARY OUTCOMES:
Changes in perceived stress scores as measured by the Perceived Stress Scale (PSS) for treatment group versus control group | Baseline, 8-weeks
  The 8-week randomized controlled trial (RCT) of the virtual chair yoga treatment versus the waitlist control group will assess the effects of the virtual chair yoga on perceived stress in older adults and caregivers, using the PSS.
  Scores on the PSS can range from 0-40, with higher scores indicating higher perceived stress.
  Hypothesis: Following participation in an 8-week RCT of the virtual chair yoga program, older adults with dementia and their caregivers will report lower perceived stress, as measured by the Perceived Stress Scale (PSS) compared to the waitlist control group.

SECONDARY OUTCOMES:
Changes in loneliness scores as measured by the 3-item UCLA Loneliness Scale for treatment group versus control group | Baseline, 8-weeks
  The 8-week randomized controlled trial (RCT) of the virtual chair yoga treatment versus the waitlist control group will assess the effects of the virtual chair yoga on perceived stress in older adults and caregivers, using the PSS.
  Scores on the UCLA Loneliness Scale can range from 3-9, with higher scores indicating higher loneliness.
  Hypothesis: Following participation in an 8-week RCT of the virtual chair yoga program, older adults with dementia and their caregivers will report less loneliness, as measured by the UCLA Loneliness Scale compared to the waitlist control group.

OTHER OUTCOMES:
Changes in caregiver burden as measured by the Zarit Burden Interview (ZBI) for treatment group versus control group | Baseline, 8-weeks
  The 8-week randomized controlled trial (RCT) of the virtual chair yoga treatment versus the waitlist control group will assess the effects of the virtual chair yoga on caregiver burden in caregivers, using the ZBI.
  Scores on the ZBI can range from 0-88, with higher scores corresponding to higher levels of burden.
  Hypothesis 1: Following participation in an 8-week RCT of the virtual chair yoga program, caregivers of older adults will report less caregiver burden, as measured by the Zarit Burden Interview (ZBI) compared to the waitlist control group.
  Hypothesis 2: Lower scores for older adults on the PHQ-9 and GAD-7 (week 8) will be associated with decreased caregiver burden following participation in an 8-week RCT of the virtual chair yoga program.
Changes in depressive symptoms as measured by the Patient Health Questionnaire-9 (PHQ-9) for treatment group versus control group | Baseline, 8-weeks
  The 8-week randomized controlled trial (RCT) of the virtual chair yoga treatment versus the waitlist control group will assess the effects of the virtual chair yoga on depressive symptoms in older adults and caregivers, using the PHQ-9.
  Scores on the PHQ-9 can range from 0-27, with higher scores indicating more severe depression.
  Hypothesis: Following participation in an 8-week RCT of the virtual chair yoga program, older adults with dementia and their caregivers will report less depressive symptoms, as measured by the Patient Health Questionnaire (PHQ-9) compared to the waitlist control group.
Changes in symptoms of anxiety as measured by the Generalized Anxiety Disorder-7 (GAD-7) scale for treatment group versus control group | Baseline, 8-weeks
  The 8-week randomized controlled trial (RCT) of the virtual chair yoga treatment versus the waitlist control group will assess the effects of the virtual chair yoga on symptoms of anxiety in older adults and caregivers, using the GAD-7.
  Scores on the GAD-7 range from 0-21, with higher scores indicating more severe anxiety.
  Hypothesis: Following participation in an 8-week RCT of the virtual chair yoga program, older adults with dementia and their caregivers will report less symptoms of anxiety, as measured by the Generalized Anxiety Disorder 7-Item Scale (GAD-7) compared to the waitlist control group.
Changes in fear of COVID-19 as measured by the Fear of COVID-19 scale (FC-19S) for treatment group versus control group | Baseline, 8-weeks
  The 8-week randomized controlled trial (RCT) of the virtual chair yoga treatment versus the waitlist control group will assess the effects of the virtual chair yoga on fear of COVID-19 in older adults and caregivers, using the FC-19S.
  Scores on the FC-19S range from 7-35, with higher scores indicating more fear of COVID-19.
  Hypothesis: Following participation in an 8-week RCT of the virtual chair yoga program, older adults with dementia and their caregivers will report less fear of COVID-19, as measured by the Fear of COVID-19 scale (FC-19S) compared to the waitlist control group.
Semi-structured interviews for the Qualitative Component | 8-weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Institute of Community and Family Psychiatry, Montreal, Quebec
  - Douglas Mental Health University Institute, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No